CLINICAL TRIAL: NCT01969500
Title: Development of a Mobile System for Self-management of Schizophrenia (SOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH100195-01
Record Dates: First submitted 2013-10-15; First posted 2013-10-25 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Self Management of Schizophrenia; SOS; Serious Mental Illness; Psychosis; Social Dysfunction; Medication Adherence; Mobile Application; EHealth; E-Health; Health Technology; mobile health; m-Health; electronic health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Medication Adherence | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Treatment as usual includes outpatient case management, linkage to services and medication monitoring.
  Interventions: Behavioral: Treatment as Usual (TAU)
- Mobile Application (Experimental): Mobile Application system designed to improve coping with psychotic symptoms, social functioning, and medication adherence.
  Interventions: Behavioral: Mobile Application

INTERVENTIONS:
Behavioral: Mobile Application
  Other Names: Self-Management of Schizophrenia (SOS); FOCUS
  Arms: Mobile Application
Behavioral: Treatment as Usual (TAU)
  Arms: Treatment as Usual

SUMMARY:
This 2-arm clinical trial piloted a mobile Self-Management of Schizophrenia (SOS) system that administers interventions targeting persistent symptoms of psychosis, social dysfunction, and medication adherence. Researchers compared an intervention arm using the SOS system and an arm receiving treatment as usual on the outcomes of change in severity of psychotic symptoms and change in social functioning.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV (Diagnostic and Statistical Manual IV) criteria for schizophrenia or schizoaffective disorder based on a chart diagnosis;
* 18 years or older;
* Prescribed oral antipsychotic medication; and
* A rating of "3" or lower on one of the three items which comprise the Domination by Symptoms factor from the Recovery Assessment Scale, indicating patient-rated need for illness self-management

Exclusion Criteria:

* Hearing, vision, or motor impairment that make it impossible to operate a smartphone or respond to prompts (determined using demonstration smartphone for screening); and
* English reading level below 4th grade (determined using the Wide Range Achievement Test - 4th Edition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — University of Washington
Locations (1):
- The Mental Health Center of Greater Manchester, Manchester, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with schizophrenia or schizoaffective disorder who were receiving services were recruited through flyers in waiting rooms and bulletin boards at treatment centers, and through referrals from clinical staff. Enrollment was open from November 2015 to July 2016.
Pre-assignment Details: N=3 enrolled participants were not assigned because N=1 did not pass a competency screener, N=1 did not meet Recovery Assessment Scale inclusion criteria, and N= 1 was no longer interested prior to completing baseline.
Groups:
- Treatment as Usual: Treatment as usual includes outpatient case management, linkage to services and medication monitoring.
  Treatment as Usual
- Mobile Application: Mobile Application system designed to improve coping with psychotic symptoms, social functioning, and medication adherence.
  Mobile Application
Period: Overall Study
Arm/Group | Treatment as Usual | Mobile Application
Started | 25 | 26
Completed | 24 | 24
Not Completed | 1 | 2
Not completed — Death | 0 | 1
Not completed — extended hospitalization | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Mobile Application | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (12.5) | 42.5 (13.4) | 42.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 20 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 22 | 24 | 46
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Beliefs about Medicines Questionnaire - General (BMQ - General) [Mean (Standard Deviation); unit: units on a scale] — The Beliefs about Medicine Questionnaire - General (BMQ - General) comprises two 4-item factors with 5-point Likert scales assessing beliefs that medicines are harmful, addictive, poisons which should not be taken continuously and that medicines are overused by doctors. Total scores range from 8-40. Higher scores indicate more negative beliefs about medicines. Population: N=1 participant in the mobile application arm did not complete the baseline assessment and is not included in analysis for all measures except ISI.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 19.96 (4.57) | 20.32 (4.36) | 20.14 (4.46)
Beliefs about Medicines Questionnaire - Specific (BMQ - Specific) [Mean (Standard Deviation); unit: units on a scale] — The Beliefs about Medicines Questionnaire - Specific (BMQ - Specific) comprises two 5-item factors with 5-point Likert scales assessing beliefs about the necessity of prescribed medication and concerns about prescribed medication based on beliefs about the danger of dependence, long-term toxicity, and the disruptive effects of medication. Total scores range from 10-50. Higher scores represent more negative beliefs about taking prescribed medication. Population: N=1 participant in the mobile application arm did not complete the baseline assessment and is not included in analysis for all measures except ISI.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 32.56 (5.24) | 32.20 (4.49) | 32.38 (4.86)
Schizophrenia Patient Activation Measure (SPAM) [Mean (Standard Deviation); unit: units on a scale] — The Schizophrenia Patient Activation Measure (SPAM) is an adaptation of the Patient Activation Measure (PAM). This measure is 14 items with 5-point Likert responses. It measures confidence in self-management and understanding of the participant's schizophrenia. Scores range from 14-70. Higher scores indicate more confidence in self-management and understanding of the participant's schizophrenia. Population: N=1 participant in the mobile application arm did not complete the baseline assessment and is not included in analysis for all measures except ISI.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 56.28 (5.73) | 57.48 (5.25) | 56.88 (5.49)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI) is a psychometric test for measuring the severity of depression with 21 questions on a 4-point scale. The scores range from 0-63. Higher scores indicate more severe depressive symptoms. Population: N=1 participant in the mobile application arm did not complete the baseline assessment and is not included in analysis for all measures except ISI.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 17.68 (10.85) | 14.12 (8.07) | 15.90 (9.46)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — Insomnia Severity Index (ISI) is a 7-item, 5-point Likert scale self-report instrument measuring the participant's perception of his or her insomnia. Scores range from 0 to 28. Higher scores indicate the participant perceives his or her insomnia as more severe.
  units on a scale | 7.56 (7.17) | 6.73 (5.68) | 7.15 (6.42)
Working Alliance Inventory (WAI) [Mean (Standard Deviation); unit: units on a scale] — The Working Alliance Inventory (WAI) is a 12-item scale with 7-point Likert responses that provides an overall measure of alliance between patients and clinical support workers. Scores can range from 12 to 84. Higher scores indicate a better alliance between the patient and the clinical support worker. Population: N=1 participant in the mobile application arm did not complete the baseline assessment and is not included in analysis for all measures except ISI.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 64.68 (12.93) | 66.28 (11.43) | 65.48 (12.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Psychotic Symptoms
Description: Severity of Psychotic Symptoms was assessed with the Psychotic Symptom Rating Scales (PSYRATS). The PSYRATS is comprised of 17 items inquiring about the specific dimensions of hallucinations and delusions, with each item being rated from 0 (absent) to 4 (severe). The PSYRATS has 2 subscales: the auditory hallucinations subscale (AHS) consisting of 11 items, and the delusions subscale (DS) consisting of 6 items. These subscale scores are added to create a total score ranging from 0-68. Higher scores indicate worse symptoms.
Time Frame: Baseline, week 12
Population: N=1 participant in the mobile application arm did not complete the baseline assessment and is not included in analysis for all measures except ISI.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment as Usual | Mobile Application
Number analyzed (Participants) | 25 | 25
units on a scale
  baseline | 20.20 (3.20) | 19.88 (3.20)
  12 weeks | 21.98 (3.24) | 20.96 (3.24)
Statistical Analysis 1: Comparison: Treatment as Usual vs Mobile Application; Test type: Superiority; p = .85, Linear mixed effects model; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-8.37 to 6.96], Standard Error of Mean 3.81 — Mean difference (Intervention Arm - TAU) in change from baseline to 12 weeks

2. Primary Outcome: Change in Social Functioning
Description: Social Functioning was measured using two subscales from the Social Functioning Scale (SFS): Social Engagement (5-items) and Withdrawal & Communication (10-items). The item values range from 0 (almost never) to 3 (often). The two subscales were summed to give a score between 0-45. A higher score indicates greater social functioning.
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment as Usual | Mobile Application
Number analyzed (Participants) | 25 | 25
units on a scale
  baseline | 27.60 (1.15) | 25.96 (1.15)
  12 weeks | 29.28 (1.17) | 26.34 (1.17)
Statistical Analysis 1: Comparison: Treatment as Usual vs Mobile Application; Test type: Superiority; p = .44, Linear mixed effects model; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-4.66 to 2.06], Standard Error of Mean 1.67 — Mean difference (Intervention Arm - TAU) in change from baseline to 12 weeks

3. Secondary Outcome: Change in System Use
Description: System use was measured by the SOS application regarding the percent of SOS prompts and self-report interactions with the system.
Time Frame: 4 weeks
Population: This data was collected in a previous field trial, not in this randomized controlled trial.
Arm/Group | Treatment as Usual | Mobile Application
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Usability and Satisfaction
Description: Usability and Satisfaction was measured using the USE (Usefulness, Satisfaction, and Ease of use) Questionnaire, which was designed to measure satisfaction, usefulness, ease of use and ease of learning.
Time Frame: 4 weeks
Population: This data was collected in a previous field trial, not in this randomized controlled trial.
Arm/Group | Treatment as Usual | Mobile Application
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed at the baseline and 12 week assessments for each participant.
Arm/Group | Treatment as Usual | Mobile Application
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT01969500/Prot_SAP_000.pdf